CLINICAL TRIAL: NCT03739749
Title: Arthroscopic Superior Capsular Reconstruction - Multicentric Prospective Comparative Study of Different Types of Grafts
Brief Title: Arthroscopic Superior Capsular Reconstruction - Study of Different Types of Grafts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Multicenter failure
Sponsor: Hospital de Egas Moniz (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government); General Hospital of Santo António (Other); Centro Hospitalar De São João, E.P.E. (Other); Hospital Santa Maria Maior de Barcelos (Unknown); CUF Santarém Hospital (Other); Hospital de Braga (Other); Unidade Local de Saúde de Coimbra, EPE (Other); Hospital Cuf Descobertas (Unknown); Hospital Vila Franca de Xira (Other)
Responsible Party: Principal Investigator, Clara Isabel de Campos Azevedo, Principal Investigator, Hospital de Egas Moniz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2018-10HSFX
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Rotator Cuff Tear; Graft Complication
Keywords: Arthroscopic Superior Capsular Reconstruction; Irreparable rotator cuff tear; Allograft; Autograft; Xenograft
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Multiple group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fascia lata autograft (Active Comparator): Arthroscopic superior capsular reconstruction using a fascia lata autograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction
- Fascia lata allograft (Active Comparator): Arthroscopic superior capsular reconstruction using a fascia lata allograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction
- Achilles tendon allograft (Active Comparator): Arthroscopic superior capsular reconstruction using an achilles tendon allograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction
- Bovine pericardium allograft (Active Comparator): Arthroscopic superior capsular reconstruction using a bovine pericardium allograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction
- Swine dermal xenograft (Active Comparator): Arthroscopic superior capsular reconstruction using a swine dermal xenograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction
- Collagen allograft (Active Comparator): Arthroscopic superior capsular reconstruction using a collagen allograft
  Interventions: Procedure: Arthroscopic superior capsular reconstruction

INTERVENTIONS:
Procedure: Arthroscopic superior capsular reconstruction — The superior capsule of patients with irreparable rotator cuff tears will be reconstructed using an autograft or an allograft

SUMMARY:
Multicentric prospective clinical and radiological comparative study of consecutive patients with irreparable rotator cuff tears to test the hypothesis that there are significant differences in the improvement of the clinical and imaging outcomes of arthroscopic superior capsular reconstruction (ASCR) when a different type of graft is used.

DETAILED DESCRIPTION:
Patients with irreparable rotator cuff tears who meet the eligibility criteria will be enrolled in the study and undergo arthroscopic superior capsular reconstruction using one of the following types of graft: fascia lata autograft, fascia lata allograft, Achilles tendon allograft, bovine pericardium xenograft, swine dermal xenograft, or collagen graft.

All patients will be assessed clinically, radiologically and with an MRI preoperatively and at the 6-months and at the 2-years postoperative evaluations. The range of motion (ROM), shoulder abduction strength, Constant (CS), simple shoulder test (SST) and subjective shoulder value (SSV) scores will be compared from preoperative to 6 months postoperative; from 6 months postoperative to 2 years postoperative (paired-samples t-test, two-tailed) in each group (allotment to groups is performed according to the type of graft used: fascia lata autograft, fascia lata allograft, Achilles tendon allograft, bovine pericardium xenograft, swine dermal xenograft, or collagen graft). The differences in ROM, shoulder abduction strength, CS, SST and SSV scores from preoperative to 6 months postoperative and from 6 months postoperative to 2 years postoperative will be compared between groups. All continuous variables will be compared between the group of patients with graft tears and the group without graft tears (Mann-Whitney U test). All categorical variables and outcome results will be compared between groups (Fisher's exact test). A significant difference will be defined as P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tear arthropathy, Hamada stage 1 or 2
* Complete rotator cuff tendon tear involving one or more tendons, with a Patte stage 3 tendon retraction on the preoperative magnetic resonance imaging

Exclusion Criteria:

* Rotator cuff tear arthropathy, Hamada stage 3 or 4
* Complete rotator cuff tendon tear involving one or more tendons, with Patte stage 1 or 2 tendon retraction on the preoperative magnetic resonance imaging
* Proximal humerus fracture
* Acute shoulder dislocation (in the previous 8 weeks)

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Constant score | 2 years
  Constant score at 2 years postoperatively (minimum 1 point - maximum 100 points); For the scale range provided, higher values represent a better outcome

SECONDARY OUTCOMES:
Graft integrity on the magnetic resonance imaging | 2 years
  Graft integrity on the 2-year postoperative magnetic resonance imaging (scale: 0 -1): 0 = graft absent or not healed to the greater tuberosity/superior glenoid; 1 = graft present and healed to the greater tuberosity and superior glenoid. For the scale range provided, higher values represent a better outcome.
Shoulder active range of motion | 2 years
  Shoulder active range of motion (ROM) at 2 years postoperatively measured in degrees using an analogic goniometer: elevation (0 - 180º), abduction (0 - 180º) and external rotation (0 - 100º); and internal rotation, defined as the highest vertebral body that the patient's thumb can reach, converted afterwards to a scale of 1 - 5 points: lateral thigh=0; buttock=1; sacrum=2; lumbar=3; 12th thoracic vertebra=4; 7th thoracic vertebra=5. For the scale range provided, higher values represent a better outcome.
Simple shoulder test | 2 years
  Simple shoulder test ((minimum 1 point - maximum 12 points) at 2 years postoperatively. For the scale range provided, higher values represent a better outcome.
Acromiohumeral interval | 2 years
  True anteroposterior shoulder radiograph at 2 years postoperatively: the acromiohumeral interval (AHI), considering the distance between the top of the humeral head and the undersurface of the acromion, measured using a software measurement tool (PACS, Agfa HealthCare); the RCT arthritis will be graded according to the Hamada revised radiographic classification. For the scale range provided, higher values represent a better outcome.
Shoulder strength | 2 years
  Shoulder strength at 2 years postoperatively measured in kilograms using a digital dynamometer: supraspinatus (0 - 25 kg).For the scale range provided, higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Azevedo, Principal Investigator — Centro Hospitalar de Lisboa Ocidental
Locations (1):
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lippitt S, Harryman DT, Matsen F. A pratical tool for function evaluation: the
- [Background] Patte D. Classification of rotator cuff lesions. Clin Orthop Relat Res. 1990 May;(254):81-6. PMID 2323151
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Gilbart MK, Gerber C. Comparison of the subjective shoulder value and the Constant score. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):717-21. doi: 10.1016/j.jse.2007.02.123. PMID 18061114